CLINICAL TRIAL: NCT07194278
Title: Feasibility and Preliminary Results of the Efficacy of Blue-Blocking Glasses on Manic Symptoms in Bipolar Disorder
Acronym: B2Bi
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier St Anne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: D24_EPI039; 2024-A00802-45 (Other: ANSM)
Record Dates: First submitted 2025-02-04; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Bipolar 1 Disorder
Keywords: bipolar 1 disorder; blue-blocking glasses; manic episode
MeSH Terms: conditions — Mania

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Groupe intervention (Experimental): he intervention will last for 7 days, during which patients are required to wear the glasses from 6 p.m. to 8 a.m. and whenever a light is turned on during this interval. Additionally, patients will be asked to wear an actimeter and fill out a sleep diary each day. Doctors will conduct daily interviews to assess manic symptoms, with more in-depth assessments scheduled on days 0, 3, and 7 to evaluate other clinical characteristics.
  Interventions: Device: Blue-blocking glasses

INTERVENTIONS:
Device: Blue-blocking glasses — The intervention will last for 7 days, during which patients are required to wear the glasses from 6 p.m. to 8 a.m. and whenever a light is turned on during this interval. Additionally, patients will be asked to wear an actimeter and fill out a sleep diary each day. Doctors will conduct daily interviews to assess manic symptoms, with more in-depth assessments scheduled on days 0, 3, and 7 to evaluate other clinical characteristics.

SUMMARY:
The goal of this clinical trial is to assess the feasibility of conducting a clinical trial of the use of blue-blocking glasses among patients with a type1 bipolar disorder, experiencing a manic episode. The feasibility criteria include: recruitment rates, participation rates, adherence to the research protocol, the material feasibility of the study. Feasibility criteria will be assessed at the end of the study period.

The investigators also want to assess patients' acceptability regarding the use of blue-blocking glasses during a manic episode, using self-reported satisfaction criteria. Those criteria will be monitored at the end of participation period for each patient (7 days after inclusion).

In addition, the study will evaluate the impact of the use of blue-blocking glasses on the severity of manic symptoms, sleeping pattern (quality of sleep, sleep latency, night wake, etc.), global functioning, and on suicidal ideations. Those indicators will be assessed at day 0 (inclusion), day 3 and day 7, using validated questionnaires and actimetry data.

The study is presented to all patients over 18 years old, with type 1 bipolar disorder, presenting a manic episode, hospitalised in an adult psychiatric ward of Bichat Hospital (GHU Paris).

Patients' participation duration is of 7 days after inclusion.

DETAILED DESCRIPTION:
1. Patients' recruitment Patients experiencing a manic episode within the context of bipolar disorder type 1 will be recruited from the hospitalization department of sector G22 at GHU-Paris, located at the Maison Blanche - Bichat site. The physicians treating eligible patients will be able to invite them to participate in the study. They will provide an information sheet and explain the aims and objectives of the study, as well as the constraints related to participation. Patients suffering from a manic episode according to DSM-5 criteria are routinely hospitalized for longer than the intervention duration (7 days). Therefore, the entire follow-up can be conducted within the hospitalization service.
2. Inclusion and study visits The participant will complete an initial questionnaire upon inclusion (D0), followed by two visits at D3 and D7 (end of the intervention). These are hetero-questionnaires to be completed via questionnaires on the RedCap® software. Additionally, participants will be asked to wear an actimetry watch continuously for the 7 days of the intervention.

   2.1) Inclusion Visit

   Once inclusion criteria are verified, the patient informed, and consent obtained, the inclusion questionnaire will be completed by the clinician in the presence of the participant. The inclusion questionnaire will consist of several sections:
   * Sociodemographic data: age, sex, year of birth, lifestyle, education level, and professional activity.
   * Clinical data: the psychiatric pathology presented by the participant, psychiatric and somatic comorbidities, ongoing medications.
   * Evaluation of addictive behaviours (tobacco, alcohol, other psychoactive substances) through frequency and consumption level.
   * Evaluation of clinical efficacy criteria based on the Young Mania Rating Scale (YMRS).
   * The participant will also complete sleep evaluation questionnaires:

     * Pittsburgh Sleep Quality Index (PSQI): a self-assessment questionnaire evaluating sleep quality; it consists of 19 questions and takes 5-10 minutes to complete.
     * Insomnia Severity Index (ISI): a short scale (7 questions) to assess the nature of insomnia, sleep satisfaction, daily functioning, and anxiety about sleep disturbances.

   During the inclusion visit, the participant will be provided with blue-blocking glasses along with the medical usage protocol and the actimetry watches. The patient will also begin filling out the sleep diary starting from inclusion.

   2.2) Follow-up visits The YMRS questionnaire will be administered daily during the intervention. The patient will complete the sleep diary every day during the intervention. Two follow-up visits are scheduled during the intervention, on D3 and D7, during which sleep evaluation questionnaires will be re-administered to the participants, and an update of ongoing medications will be performed by the clinician.

   The acceptability questionnaire will be given to the patient during the last visit (D7).

   The feasibility questionnaire will be completed at the end of the intervention (D7).

   The actimeter will be provided at inclusion with a sleep diary and will be collected at the end of the intervention on D7.
3. Data collection 3.1) Feasibility Evaluation

   Feasibility will be evaluated based on several elements related to participant recruitment, the intervention process, and the quality of the collected data. The indicators calculated are presented below in section 7.2. This evaluation will focus on the following points:
   1. Availability of the targeted population at the participating centre (number of eligible patients, number of patients who accepted participation, number of included patients);
   2. The eligibility criteria for participants, as defined in the protocol, are realistic and allow the inclusion of a sufficient number of appropriate subjects within the established recruitment period;
   3. The constraints associated with participation in the study (delivery and retrieval of study material, application of the medical procedure, number and duration of visits, etc.) have been respected, along with any reported side effects;
   4. The intervention has been conducted according to the procedure outlined in the study protocol (adherence to instructions provided to patients);
   5. The data collected via the e-CRF is complete and of high quality. Beyond these indicators, the necessary resources for conducting the clinical study at the site will also be evaluated: assessing the time dedicated by clinicians to recruit patients (presentation of the study and participation constraints, consent signing, etc.) and the personnel involved in the research (clinical study technicians, etc.).

   The investigators will also collect data on the characteristics of included patients compared to those not included, excluded, who did not consent to the research, or who withdrew prematurely from the study.

   3.2) Acceptability Evaluation Acceptability will be measured among participants using a specific questionnaire.

   The questions will focus on the level of constraint of wearing the glasses, reasons for non-compliance with instructions, the perceived usefulness of the glasses, and the level of satisfaction with using the glasses during the intervention.

   The questions are partly derived from a controlled trial by Henriksen et al., assessing the impact of blue-blocking glasses on manic symptoms in patients with bipolar disorder. The patient should evaluate their agreement with several statements (strongly disagree, somewhat disagree, neither disagree nor agree, somewhat agree, strongly agree) regarding blue-light blocking glasses comfort, burden, effective, etc. The same will apply to the actimeter watch.

   3.3) Clinical Efficacy Evaluation Clinical efficacy will be evaluated using the Young Mania Rating Scale (YMRS). This scale includes 11 items for manic symptoms: euphoria, increased activity/motor energy, sexual interest, sleep, irritability, speech (rate and amount), language disturbance, thought content, behavioural aggression/aggressiveness, appearance, and clarity. The total score is obtained by summing the scores of the 11 items. Each item is rated on a 5-point scale from 0 to 4 (from 0 - absence of symptoms to 4 - extreme symptoms). The scale interpretation is as follows: total score < 6 = euthymia, 7-20 = hypomanic episode, total score > 20 = manic episode. The scale is administered daily by a clinician during a 15-30-minute interview.

   A reduction in the severity of mania in patients from the start to the end of the intervention will support the clinical efficacy of using blue-light blocking glasses.
4. Sample size As a feasability study, 25 patients will be included, as it was done in previous similar trials.
5. Risk assessment Few side effects were reported during virtual darkness therapy within the time intervals specified in the protocol. The reported side effects are: reversible headaches, mild depressive symptoms that quickly resolve, and energy loss in the evening.

   The risk of adverse effects (AEs) related to the intervention is considered minimal, if not non-existent. Any adverse event will be reported by the investigator to the sponsor via a specific AE reporting form. In the case of a serious adverse event, the sponsor will report it to the Ethics Committee (CPP) and health authorities.

   The frequency of AEs will be monitored by the project team throughout the participant inclusion period.

   Anyone experiencing an adverse event (serious or not) will receive appropriate care based on their condition and will be followed up until the event resolves or until the end of the study. If necessary, the intervention/study will be stopped.

   The criteria for study withdrawal are:
   * By decision of the physician: deterioration in somatic or psychiatric status requiring premature cessation of study participation.
   * By decision of the participant: withdrawal from the study
   * Premature withdrawal will also be justified by the end of hospitalization or transfer to another non-participating care unit.
6. Ethical considerations The study was approved by the Comité de Protection des Personnes. The healthcare professional monitoring an eligible patient will present the study to them and provide an information sheet, along with a study booklet that outlines the study objectives and participation details. If the participant agrees, they will be invited to sign the informed consent form.

The information sheet will include the contact details of the data controller and the Data Protection Officer (DPO) for any questions related to data protection or to object to the future use of the data.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old
* Patient with a type 1 bipolar disorder presenting a manic episode according to the DSM-5 TR, with or without associated psychotic disorders.

Exclusion Criteria:

* Patient who did not agree to participate to the study
* Patient unable to be informed or understand the course of the study
* Patient with severe eye problem or with an history of trauma affecting the eyes
* Pregnant or breastfeeding women
* Patient in need of urgent care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-07-19 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Feasability | 7 days after admission
  Feasibility of the intervention will be assessed with an ad hoc questionnaire including recruitment rate, participation rate, the acceptability of the study protocol, patients' commitment to the intervention, etc.

SECONDARY OUTCOMES:
Patients' acceptability of the intervention | 7 days after admission
  Assessment is based on self-reported satisfaction criteria regarding the use of blue-blocking glasses, and to identify potential barriers to their use by bipolar patients.
Efficacy of blue-blocking glasses | Day 0, day 3 and day 7
  Efficacy of the use of blue-blocking glasses among bipolar patients experiencing a manic episode is assessed with the Young Mania Rating Scale (YMRS).
  Use as a tool to assess and record the severity of a manic episode. The questionnaire consists of eleven items which the clinician rates based on the assessment of the patients current condition during the course of the interview. The total score which ranges from 0-60. A score of 20-30 points indicate moderate mania and >30 points indicate severe mania.
Impact on sleep quality | Day 0, day 3 and day 7
  Impact on sleep quality is evaluated by the Pittsburgh Sleep Quality Index (PSQI). The global score ranges 0 to 21. Higher scores indicate worse sleep quality.
Suicidal risk | Day 0 and day 7
  Suicidal risk is determined using the Columbia Suicide Severity Rating Scale (CSSRS). It contains 6 "yes" or "no" questions to rate an individual's degree of suicidal ideation. Interpretation : 0 = No risk reported (all "no" responses) · 1 - 2 points = Low risk · 3 - 6 points = Moderate to high risk.
Global functioning | 7 days after admission
  Global functioning is evaluated by a standardised scale, Clinical Global Impression (CGI), which is rated on a 7-point scale, with the severity of illness ranging from 1 (normal) through to 7 (the most severely ill )
Impact on sleep quality | Day 0, day 3 and day 7
  Presence of insomnia will be assessed by the Insomnia Severity Index (ISI). The total score ranges from 0 to 28. Interpretation : absence of insomnia (0-7); sub-threshold insomnia (8-14); moderate insomnia (15-21); and severe insomnia (22-28).
Impact on sleep quality | Day 0, day 3 and day 7
  Sleep/wake patterns will be measured with actimetry data.

CONTACTS AND LOCATIONS:
Locations (1):
- Secteur de psychiatrie adulte G22-G23-G24, Paris, France, France

IPD SHARING:
Plan to Share IPD: Undecided
Need to consider French regulation policies